CLINICAL TRIAL: NCT00392223
Title: A Phase III, Multicenter, Randomized, Double Blind-Double Dummy Study, To Evaluate Efficacy And Safety Of Treatment With Azithromycin, Microspheres, Oral Powder For Suspension, 2 G, In One Administration A Week, For 8 Weeks, Compared With Treatment With Minocycline Capsules, 100 Mg Die For 8 Weeks, In Outpatients With Moderate To Severe Inflammatory Acne.
Brief Title: Efficacy And Safety Of Azithromycin SR Compared With Minocycline In Acne
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661150
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline

ARMS (2):
- Treatment Group A (Experimental)
  Interventions: Drug: Azithromycin microspheres; Drug: minocycline-placebo capsules
- Treatment Group B (Experimental)
  Interventions: Drug: Azithromycin microspheres-placebo; Drug: Minocycline capsules,

INTERVENTIONS:
Drug: Azithromycin microspheres — Azithromycin microspheres, powder for oral suspension, 2 g a week, in unique administration PO, repeated weekly for 8 weeks and minocycline-placebo capsules daily for 8 weeks plus minocycline placebo
  Arms: Treatment Group A
Drug: minocycline-placebo capsules — minocycline-placebo capsules daily for 8 weeks plus minocycline placebo
  Arms: Treatment Group A
Drug: Azithromycin microspheres-placebo — Minocycline capsules, PO, 100 mg daily for 8 weeks and Azithromycin microspheres-placebo once a week for 8 weeks plus azithromycin placebo.
  Arms: Treatment Group B
Drug: Minocycline capsules, — Capsules, PO, 100 mg daily for 8 weeks.
  Arms: Treatment Group B

SUMMARY:
The primary objective is to evaluate the clinical efficacy of azithromycin microspheres treatment in outpatients with moderate to severe inflammatory acne compared with first line treatment minocycline after 8 weeks of therapy

DETAILED DESCRIPTION:
The study prematurely discontinued on the February 1, 2008 due to slow enrollment.It should be noted that safety concerns have not been seen in this study and have not factored into this decision.

ELIGIBILITY:
Inclusion Criteria:

* male and female, > 16 years of age, with diagnosis of acne papulo-pustular, moderate (19-30 GAGS score) to severe (31-33 GAGS score)

Exclusion Criteria:

* pregnancy, gastrointestinal and endocrinological disease, specific systemic disease, hormonal contraceptives, isotretinoin, topic drugs for acne (except detergent allowed)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Italy (16):
  - Pfizer Investigational Site, Germona Del Friuli, Udine
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Catanzaro
  - Pfizer Investigational Site, Ferrara
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Lucca
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Pordenone
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Siena
  - Pfizer Investigational Site, Terni
  - Pfizer Investigational Site, Trieste

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661150&StudyName=Efficacy%20And%20Safety%20Of%20Azithromycin%20SR%20Compared%20With%20Minocycline%20In%20Acne%20%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: 2 grams per week administered orally (PO) for 8 weeks (azithromycin microspheres, powder for oral suspension)
- Minocycline: 100 milligrams (mg) administered PO (oral) QD (every day) for 8 weeks (minocycline capsules)
Period: Overall Study
Arm/Group | Azithromycin | Minocycline
Started | 58 | 60
Completed | 49 | 47
Not Completed | 9 | 13
Not completed — Adverse Event | 5 | 4
Not completed — Lost to Follow-up | 1 | 4
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Minocycline | Total
Number analyzed (Participants) | 58 | 60 | 118
Age, Customized [Number; unit: participants]
  <18 years | 10 | 17 | 27
  Between 18 and 44 years | 48 | 43 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment in Global Acne Grading System (GAGS) Score
Description: GAGS used to assess 6 locations on face/chest/upper back; factor for each location based on surface area, distribution, density of pilosebaceous units. Locations graded separately 0 - 4 (hi). Global score factored based on summing of local scores. Change: (Global) score at observation minus (global) score at baseline.
Time Frame: Baseline, Week 8 End of Treatment (EOT)
Population: Full Analysis Set, Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Azithromycin | Minocycline
Number analyzed (Participants) | 53 | 59
score on scale | -8.69 [-10.33 to -7.05] | -9.16 [-10.62 to -7.71]
Statistical Analysis 1: Comparison: Azithromycin vs Minocycline; Test type: Non-Inferiority or Equivalence — Analysis performed to assess non-inferiority by calculation & examination of 95% CI. Analysis conducted via analysis of covariance (ANCOVA) including corresponding baseline value and centre as covariates. Non-inferiority margin was chosen as largest clinically acceptable difference. This was set as difference of 3 in GAGS global score. Azithromycin declared non-inferior to minocycline when two-sided 95% confidence interval for difference lied entirely to right of non-inferiority margin; Mean Difference (Final Values) = -0.47, 95% CI [-2.48 to 1.54] — Comparison between treatment groups was performed using an analysis of covariance (ANCOVA) method, with treatment, center, and baseline value GAGS global score included as covariates

2. Secondary Outcome: Change From Baseline in Global Acne Grading System (GAGS) Score
Description: GAGS used to assess 6 locations on face/chest/upper back; factor for each location based on surface area, distribution, density of pilosebaceous units. Locations graded separately 0 - 4 (hi. Global score factored based on summing of local scores. Change: mean at observation minus baseline.
Time Frame: Baseline, Week 4, Week 8 End of Treatment (EOT), 8 weeks after EOT
Population: Full Analysis Set. Where noted: LOCF = Last Observation Carried Forward technique was used. Number of subjects with analyzable data: n=azithromycin, minocycline (respectively).
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Azithromycin | Minocycline
Number analyzed (Participants) | 53 | 59
score on scale
  Week 4 (n=50,56) | -7.0 (7.05) [-8.33 to -5.59] | -6.5 (6.45) [-7.77 to -5.16]
  Week 8 EOT (End of Treatment) (n=52,56) | -9.7 [-11.66 to -7.77] | -10.2 [-11.86 to -8.57]
  Week 8 EOT (LOCF) (n=53,59) | -9.5 [-11.47 to -7.59] | -9.8 [-11.48 to -8.12]
  8 weeks after EOT (n=49,49) | -11.1 [-13.42 to -8.82] | -12.9 [-14.79 to -11.01]

3. Post Hoc Outcome: Number of Subjects With Mild, Moderate, and Severe Acne
Description: Global Acne Grading System score used to assess 6 locations on face/chest/upper back; factor for each based on area, distribution, density of pilosebaceous units. Locations graded separately 0 - 4 (hi). Global score factored based on sum of local scores and se verity: 0=no acne, 1-18=mild, 19-30=moderate, 31-38=severe, >39=very severe.
Time Frame: Baseline, Week 8 End of Treatment (EOT)
Population: Full Analysis Set. Where noted: LOCF = Last Observation Carried Forward technique was used.
Measure: Number; unit: participants
Arm/Group | Azithromycin | Minocycline
Number analyzed (Participants) | 53 | 59
participants
  Baseline Mild acne | 0 | 1
  Baseline Moderate acne | 49 | 52
  Baseline Severe acne | 3 | 5
  Baseline Very severe acne | 1 | 1
  Baseline Missing | 0 | 0
  Week 8 EOT (LOCF) Mild acne | 31 | 41
  Week 8 EOT (LOCF) Moderate acne | 19 | 16
  Week 8 EOT (LOCF) Severe acne | 1 | 0
  Week 8 EOT (LOCF) Very severe acne | 0 | 1
  Week 8 EOT (LOCF) Missing | 2 | 1

4. Secondary Outcome: Improvement of Global Acne Grading System (GAGS) Score
Description: Number of subjects by improvement category of GAGS score: Best improvement = reduction of GAGS score >75% (pre-post evaluation); Good improvement = reduction score > 50 - 75%; Moderate improvement : reduction score > 25 - 50%; Light improvement : reduction score > 0 - 25%; No change = reduction score = 0%; Worsening = increase score > 0 %.
Time Frame: Week 4, Week 8 End of Treatment (EOT), 8 weeks after EOT
Population: Full Analysis Set. Where noted: LOCF = Last Observation Carried Forward technique was used.
Measure: Number; unit: participants
Arm/Group | Azithromycin | Minocycline
Number analyzed (Participants) | 53 | 59
participants
  Week 4 Best Improvement | 1 | 1
  Week 4 Good Improvement | 4 | 2
  Week 4 Moderate Improvement | 19 | 25
  Week 4 Light Improvement | 23 | 24
  Week 4 No Change | 2 | 2
  Week 4 Worsening | 1 | 2
  Week 4 Missing | 3 | 3
  Week 8 EOT Best Improvement | 4 | 3
  Week 8 EOT Good Improvement | 11 | 16
  Week 8 EOT Moderate Improvement | 21 | 20
  Week 8 EOT Light Improvement | 11 | 15
  Week 8 EOT No Change | 2 | 2
  Week 8 EOT Worsening | 3 | 0
  Week 8 EOT Missing | 1 | 3
  Week 8 EOT LOCF Best Improvement | 4 | 3
  Week 8 EOT LOCF Good Improvement | 11 | 16
  Week 8 EOT LOCF Moderate Improvement | 21 | 20
  Week 8 EOT LOCF Light Improvement | 11 | 17
  Week 8 EOT LOCF No Change | 3 | 2
  Week 8 EOT LOCF Worsening | 3 | 1
  Week 8 EOT LOCF Missing | 0 | 0
  8 weeks after EOT Best Improvement | 7 | 6
  8 weeks after EOT Good Improvement | 15 | 17
  8 weeks after EOT Moderate Improvement | 13 | 18
  8 weeks after EOT Light Improvement | 6 | 8
  8 weeks after EOT No Change | 3 | 0
  8 weeks after EOT Worsening | 5 | 0
  8 weeks after EOT Missing | 4 | 10

5. Primary Outcome: Change From Baseline to End of Treatment (EOT) in Global Acne Grading System (GAGS) Score - Per Protocol Population
Description: as for outcome 1
Time Frame: Baseline, Week 8 EOT
Population: Per Protocol population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Azithromycin | Minocycline
Number analyzed (Participants) | 48 | 48
score on scale | -9.35 [-10.75 to -7.94] | -10.22 [-11.54 to -8.90]
Statistical Analysis 1: Comparison: Azithromycin vs Minocycline; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.87, 95% CI [-2.58 to 0.84] — ANCOVA adjusted for baseline, center and treatment

6. Secondary Outcome: Change From Baseline in Acne Graded by Leeds Technique
Description: Leeds Grading technique: evaluates three sites (face, back, chest) on a 0 to 10 grading scale where 0 equals to no acne and 10 equals to most severe acne.
Time Frame: Baseline, Week 4, Week 8 End of Treatment (EOT), 8 weeks after EOT
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on scale
Arm/Group | Azithromycin | Minocycline
Number analyzed (Participants) | 53 | 59
score on scale
  Face Week 4 (n=50, 56) | -1.5 [-1.82 to -1.14] | -1.3 [-1.60 to -1.05]
  Face Week 8 EOT (n=52, 56) | -2.5 [-3.06 to -2.01] | -2.4 [-2.84 to -2.02]
  Face Week 8 EOT (LOCF) (n=53,59) | -2.5 [-3.01 to -1.97] | -2.3 [-2.74 to -1.91]
  Face 8 weeks after EOT (n=49,49) | -3.0 [-3.65 to -2.35] | -2.9 [-3.44 to -2.39]
  Back Week 4 (n=50,56) | -1.1 [-1.58 to -0.70] | -0.9 [-1.21 to -0.61]
  Back Week 8 EOT (n=52,56) | -1.5 [-1.98 to -1.02] | -1.4 [-1.83 to -1.06]
  Back Week 8 EOT (LOCF) (n=53,59) | -1.5 [-1.96 to -1.02] | -1.4 [-1.76 to -0.99]
  Back 8 weeks after EOT (n=49,49) | -1.5 [-2.03 to -0.95] | -2.0 [-2.52 to -1.40]
  Chest Week 4 (n=50,56) | -0.8 [-1.12 to -0.48] | -0.7 [-0.99 to -0.40]
  Chest Week 8 EOT (n=52,56) | -1.5 [-2.04 to -0.92] | -1.2 [-1.57 to -0.75]
  Chest Week 8 EOT (LOCF) (n=53,59) | -1.5 [-2.00 to -0.90] | -1.1 [-1.51 to -0.73]
  Chest 8 weeks after EOT (n=49,49) | -1.5 [-2.10 to -0.92] | -1.8 [-2.32 to -1.23]

ADVERSE EVENTS:
Arm/Group | Azithromycin | Minocycline
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 29 | 21
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Azithromycin | Minocycline
Eyelid edema (Eye disorders) | 0/58 | 1/60
Abdominal pain (Gastrointestinal disorders) | 7/58 | 3/60
Abdominal pain, upper (Gastrointestinal disorders) | 5/58 | 2/60
Constipation (Gastrointestinal disorders) | 1/58 | 0/60
Diarrhea (Gastrointestinal disorders) | 10/58 | 2/60
Gastritis (Gastrointestinal disorders) | 2/58 | 1/60
Gastrointestinal disorder (Gastrointestinal disorders) | 1/58 | 0/60
Nausea (Gastrointestinal disorders) | 5/58 | 1/60
Vomiting (Gastrointestinal disorders) | 5/58 | 2/60
Fatigue (General disorders) | 1/58 | 0/60
Malaise (General disorders) | 2/58 | 0/60
Pyrexia (General disorders) | 2/58 | 4/60
Hypersensitivity (Immune system disorders) | 0/58 | 2/60
Furnucle (Infections and infestations) | 1/58 | 0/60
Influenza (Infections and infestations) | 1/58 | 1/60
Localized infection (Infections and infestations) | 0/58 | 1/60
Nasopharyngitis (Infections and infestations) | 2/58 | 2/60
Otitis media acute (Infections and infestations) | 0/58 | 1/60
Pharyngitis (Infections and infestations) | 0/58 | 2/60
Tonsillitis (Infections and infestations) | 1/58 | 1/60
Joint dislocation (Injury, poisoning and procedural complications) | 0/58 | 1/60
Alanine aminotransferase increased (Investigations) | 0/58 | 2/60
Anorexia (Metabolism and nutrition disorders) | 1/58 | 0/60
Disturbance in attention (Nervous system disorders) | 1/58 | 0/60
Headache (Nervous system disorders) | 1/58 | 3/60
Migraine (Reproductive system and breast disorders) | 0/58 | 1/60
Dysmenorrhea (Reproductive system and breast disorders) | 0/58 | 1/60
Rash (Skin and subcutaneous tissue disorders) | 0/58 | 1/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.